CLINICAL TRIAL: NCT00538018
Title: Telithromycin, Treating Adult Outpatients With Mild to Moderate Community-acquired Pneumonia (CAP) in High Bacterial Resistance Areas
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HMR3647A_4015
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Pneumonia
MeSH Terms: conditions — Pneumonia | interventions — telithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Telithromycin

SUMMARY:
Demonstrate efficacy of telithromycin over single-agent oral antibiotics usually prescribed by local guidelines ("usual care") for treating adult outpatients with mild to moderate community-acquired pneumonia (CAP) in high bacterial resistance areas.

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients with mild to moderate CAP. Diagnosis of CAP was based on the presence of fever and/or hyperleucocytosis and the new and sudden onset of at least two clinical signs and symptoms of pneumonia (cough, dyspnea or tachypnea, chills, pleuritic chest pain, purulent sputum or change in sputum character, auscultatory findings). Clinical diagnosis of CAP had to be confirmed by chest X-ray findings (e.g. presence of presumably new infiltrate). Specimens for microbiological documentation had to be collected within 24 hours prior to enrollment.

Exclusion Criteria:

* Subjects requiring parenteral antibiotic treatment.
* Subjects with severe CAP requiring hospitalization. The CAP was to be considered as severe in the presence of any of the following conditions:
* chest X-ray showing a multilobar consolidation (> 1 lobe)3 and/ or an increase in the size of the opacity by greater than or = to 50% within 48 hours of the current evaluation
* shock
* altered mental status (disorientation to person, place or time that is not known to be chronic, lethargy, stupor or coma)
* total peripheral white blood cell count < 4,000/mm3
* requirement for mechanical ventilation
* requirement for vasopressors
* acute renal failure

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 978 (Actual)
Dates: Start 2003-01; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
To compare the effect of telithromycin versus "usual care" on the total symptoms score of pneumonia and on health outcomes, in CAP adult outpatients at the end of therapy visit. | (Days 8-11)

SECONDARY OUTCOMES:
For health outcomes at the test of cure visit; e.g. additional LRTI-related antibiotic use, LRTI related hospitalization with length of stay and LRTI related office visit/emergency room visit. | (Days 17-21)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi